CLINICAL TRIAL: NCT02074436
Title: Randomized Trial of Epsilon Aminocaproic Acid Versus Platelet Transfusions for the Prevention of Bleeding in Thrombocytopenic Patients With Hematological Malignancies
Brief Title: PRevention Of BLeeding in hEmatological Malignancies With Antifibrinolytic (Epsilon Aminocaproic Acid)
Acronym: PROBLEMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ana G. Antun, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00066504; Winship2429-13 (Other: Winship Cancer Institute/Emory University)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Hematological Malignancies; Thrombocytopenia
Keywords: hematological malignancies; thrombocytopenia; aminocaproic acid
MeSH Terms: conditions — Hematologic Neoplasms; Thrombocytopenia | interventions — Aminocaproic Acid; Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic EACA (Experimental): Prophylactic EACA 1000 mg PO twice daily if platelets < 20 x 10⁹/L
  Interventions: Drug: EACA
- Platelet transfusion (Active Comparator): Platelet transfusion if platelet count is < 20 x 10⁹/L in the outpatient or < 10 x 10⁹/L in the inpatient setting
  Interventions: Other: Platelet transfusion

INTERVENTIONS:
Drug: EACA — EACA 1000 mg twice a day. Patients will receive platelet transfusion in case of grade ≥ 2 bleeding.
  Other Names: Amicar; Aminocaproic acid
  Arms: Prophylactic EACA
Other: Platelet transfusion — Prophylactic platelet transfusion. Additional platelet transfusions will be administered in case of grade ≥ 2 bleeding.
  Arms: Platelet transfusion

SUMMARY:
STUDY BACKGROUND AND PURPOSE:

Patients with hematological malignancies (blood-related cancers) often develop thrombocytopenia (low platelet count), which can be made worse by cancer treatment.

Preventive (prophylactic) platelet transfusion remains the standard of care for thrombocytopenic patients. However, bleeding remains a significant problem in these patients, affecting approximately 20% of patients with acute myeloid leukemia and 34-58% of hematopoietic stem cell transplant recipients. Platelet transfusion refractoriness, the repeated failure to obtain satisfactory response to platelet transfusions, is a common problem. Alternatives to platelet transfusions are desperately needed for these patients.

Epsilon aminocaproic acid (EACA) blocks a process called fibrinolysis that is an essential step in the bleeding process. EACA is approved by the FDA for the treatment of severe bleeding-related diseases and complications. A small study has shown EACA to be well tolerated and associated with low risk of bleeding in patients with hematological malignancies.

This study will compare EACA versus standard prophylactic platelet transfusion for the prevention of bleeding in thrombocytopenic patients with hematological malignancies.

STUDY DESCRIPTION:

This is Phase II study to compare EACA versus standard prophylactic platelet transfusion to prevent bleeding in thrombocytopenic patients with hematological malignancies. Patients who are eligible to take part must give their written agreement before they can be enrolled.

The study will enroll 100 patients who will be assigned randomly to take EACA twice daily or to undergo standard prophylactic platelet transfusion. Patients will be followed for any bleeding events, need for platelet transfusion, and any side effects experienced. Patients will complete questionnaires to assess their quality of life while on the study.

DETAILED DESCRIPTION:
Study Treatments: Epsilon aminocaproic acid (EACA) vs. standard prophylactic platelet transfusions.

Study Title: Randomized Trial of Epsilon Aminocaproic Acid versus Platelet Transfusions for the Prevention of Bleeding in Thrombocytopenic Patients with Hematological Malignancies. (PROBLEMA trial: PRevention Of BLeeding in hEmatological Malignancies with Antifibrinolytic agents (epsilon aminocaproic acid).

Phase: Randomized Phase 2

Eligible Population: Adult patients with acute or chronic thrombocytopenia in the setting of hematological malignancies.

Summary and Study Rationale: Compare EACA to standard prophylactic platelet transfusion for the prevention of bleeding in thrombocytopenic patients with hematological malignancies.

Study Design: prospective, randomized, controlled trial.

Study Endpoints: The primary endpoint is to compare the proportion of patients who develop major (grades 3-4) bleeding in each arm.

Diagnosis and Main Inclusion Criteria: Age > 18 with hematological malignancies. Acute or chronic thrombocytopenia with platelet counts < 20 x 10⁹/L.

Number of Patients: 100 patients, 50 patients in each arm

Duration of Patient Participation: 6 months

Approximate Duration of Study: 3 years

Dosage and Administration:1,000 mg twice a day orally

Prohibited Medications/Treatment: Hydroxyurea and procoagulant agents including DDAVP, recombinant Factor VII or prothrombin complex concentrate are prohibited in patients receiving EACA.

Safety Evaluations: Clinical assessment once weekly during the first 30 days and then monthly for 6 months, complete blood count and bleeding score twice weekly the first 30 days, and then according to standard of care or at discretion of treating physician.

Statistical Analysis

* Population Analysis

  * Intention to treat (ITT) population: The ITT population includes all patients who are randomized to the study. Patients will be stratified and analyzed according to the treatment to which they were assigned.
  * Safety Population: The safety population includes all patients who have received at least 1 dose of EACA. Patients included in the safety population will be analyzed according to the treatment they received.
  * Per-protocol Population: The per-protocol population includes all patients who are randomized, receive at least one dose of study drug, and have no major protocol violations that could be expected to impact response data.
* Study Endpoints

  * Primary Endpoint: is to compare at the end of the study, the proportion of patients with major bleeding during the study period among patients randomized to receive either EACA or standard of care prophylactic platelet transfusions.
  * Secondary Endpoints include:

    * Proportion of patients with any bleeding during the study period in each arm
    * The total number of units of platelets transfused in each arm at the end of the study
    * Quality of life as measured in each arm before the study and at the end of the study
    * Safety in each arm
* Sample Size: This randomized, open-label phase II study is designed to compare the proportion of patient with major bleeding ever noted during the study. Patients will be assigned to receive prophylactic EACA (experimental arm) or prophylactic platelet (standard of care) in a 1:1 fashion. Previous studies suggest that the proportions of patients with major bleeding will be expected to be 8% and 30% in experimental arm and standard of care arm, respectively. With one sided Fisher's exact test, the sample size of 45 patients in each arm will achieve a power of 80% at the significance level of 5% to test whether prophylactic EACA can prevent major bleeding better than the standard of care. After adjusting for a 10% drop out rate, the actual required sample size will be 50 patients per arm. Therefore, the total sample size of the study will be 100 patients.
* Efficacy Analysis

  * Primary Endpoint Analysis will be performed using a one-sided Fisher's exact test to compare the proportions of patients with major bleeding during the whole study between the two arms. The significance level is set at 0.05. This primary analysis will be based on the ITT population.
  * Secondary Endpoint Analysis: one-sided t-test will be used to compare the total number of any bleeding episode noted during the study between the two arms. Two-sided t-test will be employed to compare the total number of units of platelets transfused at the end of the study between the two arms. Appropriate statistical tests (Chi-square test, t-test, Wilcoxon's rank sum test, etc.) will be conducted to compare the each score of the quality of life between the two arms before the study and at the end of the study, respectively. The change of each score of the quality of life from before the study to the end of the study will also be compared between the two arms. The safety in each arm will be also compared with Fisher's exact test. The analyses of secondary endpoints will be performed on the ITT population and the significance level will be kept at 0.05 for all tests.
* Safety Analysis: All patients receiving at least 1 dose of study drug will be considered evaluable for safety. Patients will be analyzed for safety according to the treatment which they received. Listings of laboratory test results will also be generated, and descriptive statistics summarizing the changes in laboratory tests over time will be presented. Exposure to study drug over time will also be summarized. The adverse events incidence rates, as well as the frequency of occurrence of overall toxicity, categorized by toxicity grades (severity) will be described for each treatment arm and be compared between two arms using two-sided Chi-square test or t-test.
* Quality of Life Analysis: Quality of life and health outcomes measures are being collected using EuroQoL instruments before the study and at the end of the study. Means and medians of raw scores of these questionnaires will be summarized for each treatment group for each domain and be compared between the two arms with t-test or Wilcoxon ranks sum test.
* Interim Analysis: Three interim analyses are planned after 11 patients in each arm have been randomized and their results have been obtained. Each interim analysis will focus on the primary endpoint, the proportion of patients with major bleeding ever noted during the study. To maintain an overall Type I error rate of 0.05 (1-sided), an O'Brien Fleming approach will be used which requires a 1-sided p-value < 0.001 at the first interim analysis (at 25% of total sample size). If this boundary is not crossed, then the study will continue and the second interim analysis will be conducted at 50% of the total sample side which requires a 1-sided significance level of 0.004. If this boundary is not crossed at the second interim analysis then, the study will continue and a third interim analysis will be conducted at 75% of the total sample side which requires a 1-sided significance level of 0.019. If this boundary is not crossed, the final primary analysis will be performed after completing 100% of the sample size using a 0.043 one-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 with a hematological malignancy
* Informed consent
* Thrombocytopenia with untransfused platelet counts < 20 x 10⁹/L in the out-patient or in the in-patient setting and one of the following criteria:

  * Acute thrombocytopenia in patients with hematological malignancies who are in remission and are receiving myelosuppressive consolidation chemotherapy that is expected to induce marrow aplasia for at least 2 weeks; or
  * Acute or chronic thrombocytopenia in patients with acute leukemia (myeloblastic or lymphoblastic) receiving induction or re-induction chemotherapy that is expected to induce marrow aplasia for at least 2 weeks; or
  * Expected chronic thrombocytopenia in patients with newly diagnosed marrow failure syndromes, myelodysplastic syndromes, aplastic anemia, chronic myelomonocytic leukemia or myelofibrosis; or
  * Expected chronic thrombocytopenia in patients with relapsed or refractory hematological malignancies; or
  * Hematopoietic stem cell transplant recipients with chronic thrombocytopenia due to chronic graft-versus-host disease (GVHD) or other causes

Exclusion Criteria:

* Acute promyelocytic leukemia
* Patient receiving anticoagulation
* Patient receiving antiplatelet agents
* Patient treated with antifibrinolytic agents (including EACA) within 14 days prior to screening
* Subjects receiving procoagulant agent including DDAVP, recombinant factor VII or prothrombin complex concentrate within 24 hours of enrollment
* Subject with known congenital bleeding disorders or platelet dysfunction
* Disseminated intravascular coagulation
* Fibrinogen level < 150 mg/dl
* Patients with known lupus anticoagulant or positive antiphospholipid antibody
* History of arterial or venous thromboembolic disease 6 months prior to screening
* Patient requiring platelet transfusion threshold of > 20 x 10⁹/L
* Active grade ≥ 2 bleeding at the time of randomization, including hematuria
* History of grade 4 bleeding
* Hematopoietic stem cell transplant recipient within 100 days post-transplant
* Pregnancy
* Known allergy to EACA
* History of veno-occlusive disease of the liver
* Myocardial infarction 6 months prior to screening
* Unstable angina
* Grade 2 renal dysfunction: creatinine > 2-3 times the upper limit of normal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana G. Antun, MD, MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

REFERENCES:
- [Background] Heddle NM, Cook RJ, Sigouin C, Slichter SJ, Murphy M, Rebulla P; BEST Collaborative (Biomedical Excellence for Safer Transfusion). A descriptive analysis of international transfusion practice and bleeding outcomes in patients with acute leukemia. Transfusion. 2006 Jun;46(6):903-11. doi: 10.1111/j.1537-2995.2006.00822.x. PMID 16734806
- [Background] 2. Gernsheimer, TB Platelet transfusion in the 21st century, ISBT 2011;6: 245-248
- [Background] Rebulla P, Finazzi G, Marangoni F, Avvisati G, Gugliotta L, Tognoni G, Barbui T, Mandelli F, Sirchia G. The threshold for prophylactic platelet transfusions in adults with acute myeloid leukemia. Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto. N Engl J Med. 1997 Dec 25;337(26):1870-5. doi: 10.1056/NEJM199712253372602. PMID 9407153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prophylactic EACA | Platelet Transfusion
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic EACA | Platelet Transfusion | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 20
  >=65 years | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Develop Major Bleeding Episodes
Description: The primary objective of this study is to compare the percentage of patients who develop major bleeding episodes (WHO grades 3-4) in the group randomized to receive prophylactic EACA versus standard of care prophylactic platelet transfusions.
  Grade 3 bleeding is defined as a bleed that significantly limits the patient's ability to perform routine activities despite symptomatic therapy and leads to reduction of the dose or discontinuation of the study drug.
  Grade 4 bleeding is a life-threatening bleed that requires discontinuation of the study drug and the patient is at immediate risk of death
Time Frame: 6 months
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic EACA | Platelet Transfusion
Number analyzed (Participants) | 11 | 11
Participants
  Grade 3 Bleeding | 0 | 11
  Grade 4 Bleeding | 11 | 0
Statistical Analysis 1: Comparison: Prophylactic EACA vs Platelet Transfusion; The results are from the first and only interim analysis focusing on the primary endpoint: proportion of patient with major bleeding (Grade 3 and 4) during the study. The interim analysis was performed after 11 patients in each arm were randomized and results were obtained. One-sided fisher's exact test was employed in the analysis. The null hypothesis is the probability of occurring major bleeding is the same for Arm A and Arm B; Test type: Other; p = 0.5, Fisher Exact

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Arm/Group | Prophylactic EACA | Platelet Transfusion
All-Cause Mortality (participants affected / at risk) | 5/15 | 5/14
Serious Adverse Events (participants affected / at risk) | 9/15 | 8/14
Other Adverse Events (participants affected / at risk) | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic EACA (N=15) | Platelet Transfusion (N=14)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Cardiac disorders) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Transfusion reaction (Immune system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Failure to Thrive (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic EACA (N=15) | Platelet Transfusion (N=14)
Chest Pain (Cardiac disorders) | 1 (2) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (2)
Hypotension (Cardiac disorders) | 2 (2) | 2 (2)
Lower extremity Edema (Cardiac disorders) | 5 (5) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Neutropenic Fever (Infections and infestations) | 3 (4) | 6 (7)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Mucositis (Infections and infestations) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 4 (17) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Oral Bleeding (Blood and lymphatic system disorders) | 8 (18) | 2 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1)
Subconjunctival Hemorrhage (Eye disorders) | 1 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (8)
Liver enzymes (Gastrointestinal disorders) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Confusion (Nervous system disorders) | 2 (3) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (3)
Hypokalemia (Endocrine disorders) | 5 (5) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (6) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
chills (General disorders) | 1 (1) | 3 (3)
Anorexia (General disorders) | 3 (3) | 2 (2)
Dehydration (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 5 (9) | 7 (8)
Hiccups (General disorders) | 0 (0) | 2 (2)
Low grade fever (General disorders) | 2 (2) | 2 (2)
Generalized weakness (General disorders) | 3 (3) | 1 (1)
Weight loss (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study because of recruitment difficulties lead to insufficient data collection and analysis of primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02074436/Prot_000.pdf